CLINICAL TRIAL: NCT05786690
Title: The Effect of Microprocessor Controlled Prostheses on Walking Pattern and Energy Consumption in Above Knee Ampute Patients
Brief Title: The Effect of Microprocessor Controlled Prostheses on Walking Pattern and Energy Consumption
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associated Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 34
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Amputation, Traumatic; Gait
MeSH Terms: conditions — Amputation, Traumatic | interventions — Methods; Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 17 patients with MIC prosthesis,
  Interventions: Other: Interventions
- Group 2: 17 patients with non-MIC prosthesis,
  Interventions: Other: Interventions

INTERVENTIONS:
Other: Interventions — the temporospatial and kinematic gait characteristics
  Other Names: Gait analysis

SUMMARY:
The aim of this study was to investigate MIC and non-MIC prostheses in terms of gait pattern and energy consumption in above-the-knee amputee patients.

DETAILED DESCRIPTION:
Background: The use of microprocessor controlled (MIC) prostheses has increased in recent years, but the number of studies on gait pattern and energy consumption in above-the-knee amputee patients is very low.

Objective: The aim of this study was to investigate MIC and non-MIC prostheses in terms of gait pattern and energy consumption in above-the-knee amputee patients.

Methods: This observational clinical study included 34 unilateral above-the-knee amputees, separated into two groups as Group 1 (n:17) using MIC prosthesis, and Group 2 (n:17) using non-MIC prosthesis. The patients were compared in terms of gait pattern, gait capacity, energy consumption, mobility, quality of life, and prosthesis satisfaction levels according to the type of prosthesis. 3D gait analysis, exercise tolerance test, Short Form 36 (SF-36) Health Survey Questionnaire, Locomotor Capabilities Index-5 (LCI-5), Satisfaction with Prosthesis Questionnaire (SAT-PRO) and six-minute walk test (6MWT) were used as evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

* as voluntary participation in the study
* age ≥18 years
* having a unilateral above-the-knee amputation
* the ability of independent ambulation in the community
* at least 6 months since the amputation
* use of the current prosthesis for at least 8 weeks

Exclusion Criteria:

* unwillingness to participate in the study
* age <18 years
* limb length discrepancy of ≥2 cm
* the presence of contracture or deformity
* additional amputation
* neuromuscular disease or comorbidity that may interfere with the study follow-up period of < 6 months since the amputation
* use of the current prosthesis for < 8 weeks
* being uncooperative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lower limb amputation
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2023-03-23 (Estimated); Primary Completion 2023-05-23 (Estimated); Study Completion 2023-06-02 (Estimated)

PRIMARY OUTCOMES:
6MWT | through study completion, an average of one and a half months
  6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Demir, Assoc. Prof., Principal Investigator — Gaziler PMR ER Hospital Ankara Turkiye